CLINICAL TRIAL: NCT02402855
Title: Impact of Conditional Financial Support on Pregnancy Outcomes in Pregnant Women With Low Incomes: Pragmatic Randomized Cluster Trial, With Parallel Arms
Brief Title: NAITRE (PreNAtal Care in deprIvaTed enviRonnEment)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BARDOU PREPS 2014
Record Dates: First submitted 2015-03-17; First posted 2015-03-30 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy
Keywords: Couverture Maladie Universelle; Couverture Maladie Universelle-Complémentaire; free health care
MeSH Terms: interventions — Interviews as Topic

ARMS (2):
- Group Intervention: Financial support (Experimental)
  Interventions: Other: Delivery of a prepaid payment card; Other: Interview with a sociologist
- Group Control: no financial support (Active Comparator)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Delivery of a prepaid payment card — Delivery of a prepaid payment card credited according to consultations attended
  Arms: Group Intervention: Financial support
Other: Interview with a sociologist — For a sub-group of 40 womens
  Arms: Group Intervention: Financial support
Other: No intervention
  Arms: Group Control: no financial support

SUMMARY:
This study aims to evaluate the impact of financial support on improving the management of prenatal care in pregnant women with low incomes. The judgment criterion is clinically pertinent: complications of pregnancy. This study also aims to evaluate attitudes to this approach through a qualitative survey.

It is planned to include 4000 women distributed into two arms of 2000 each. One group will receive financial support (prepaid payment card credited for each consultation attended according to the scheduled follow-up as recommended by the Haute Autorité de Santé); the other group will not. The management of the pregnancy for both groups will not be modified.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age > 18 years
* 1st consultation before the 26th week of amenorrhea
* Recipient of free health care (Couverture Maladie Universelle, Couverture Maladie Universelle-Complémentaire)
* Who have provided written informed consent to take part in the study

Exclusion Criteria:

* Persons without national health insurance cover
* Persons unable to understand the information on the study, despite the help of a translator or a person of trust if necessary
* Persons under guardianship

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 3787 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Occurence of complication(s) of pregnancy, wether maternal, fetal or neonatal | Participants will be followed for the duration of hospital stay and for a maximum of one month after the term date.

SECONDARY OUTCOMES:
Neonatal morbidity, mortality and rate of transfer of the newborn to a neonatal care unit. | Participants will be followed for the duration of hospital stay and for a maximum of one month after the term date.
  A composite outcome measure consisting of multiple measures: neonatal morbidity, mortality and rate of tranfer of the newborn to a neonatal care unit

OTHER OUTCOMES:
Maternal morbidity, mortality and rate of caesarean sections | Participants will be followed for the duration of hospital stay and for a maximum of one month after the term date.
  A composite outcome measure consisting of multiple measures: maternal mobidity, mortality and rate og caesarean sections
Number of scheduled consultations attended in agreement with the minimal follow-up recommendations of the Haute Autorité de Santé | Participants will be followed for the duration of hospital stay and for a maximum of one month after the term date.
Interview with a sociologist to evaluate perception of the intervention and evaluation of its perceived impact in follow-up of the pregnancy | About 6 weeks after delivery
Differential cost-effectiveness ratio associated with the financial support compared with the absence of support and expressed in terms of cost per complication avoided | Participants will be followed for the duration of hospital stay and for a maximum of one month after the term date.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHRU de BESANCON, Besançon
  - CHRU de BREST, Brest
  - CHU de DIJON, Dijon
  - APHP maternité Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHRU de LILLE, Lille
  - APHM Hôpital Nord, Marseille
  - APHP Hopital Robert Debré, Paris
  - Chu Saint Etienne, Saint-Etienne
  - Chu Tours, Tours

REFERENCES:
- [Derived] Bardou M, Meunier-Beillard N, Godard-Marceau A, Deruelle P, Virtos C, Eckman-Lacroix A, Debras E, Schmitz T; NAITRE Study group. Women and health professionals' perspectives on a conditional cash transfer programme to improve pregnancy follow-up: a qualitative analysis of the NAITRE randomised controlled study. BMJ Open. 2023 Mar 29;13(3):e067066. doi: 10.1136/bmjopen-2022-067066. PMID 36990483
- [Derived] Bardou M, Crepon B, Bertaux AC, Godard-Marceaux A, Eckman-Lacroix A, Thellier E, Falchier F, Deruelle P, Doret M, Carcopino-Tusoli X, Schmitz T, Barjat T, Morin M, Perrotin F, Hatem G, Deneux-Tharaux C, Fournel I, Laforet L, Meunier-Beillard N, Duflo E, Le Ray I; NAITRE Study Group. NAITRE study on the impact of conditional cash transfer on poor pregnancy outcomes in underprivileged women: protocol for a nationwide pragmatic cluster-randomised superiority clinical trial in France. BMJ Open. 2017 Oct 30;7(10):e017321. doi: 10.1136/bmjopen-2017-017321. PMID 29084796